CLINICAL TRIAL: NCT01550835
Title: Impact of Aspiration Thrombectomy During Carotid Stenting on New Ischemic Lesions Identified by Diffusion-Weighted Magnetic Resonance Imaging
Brief Title: Impact of Aspiration Thrombectomy During Carotid Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fogarty Clinical Research Inc. (Other)
Collaborators: Abbott Medical Devices (Industry); Helen Kay Foundation (Unknown); Northern Michigan Hospital Foundation's Louis A. and Sally Cannon (Unknown)
Responsible Party: Principal Investigator, James Joye, Chief Medical Officer, Fogarty Clinical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EV-10322
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Carotid Artery Stenosis
Keywords: Symptomatic carotid artery stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distal Embolic Protection Only (Experimental): Carotid stenting with distal embolic protection only
  Interventions: Device: Emboshield NAV6® embolic protection system (Abbott Vascular, Santa Clara, CA)
- Distal embolic protection and aspiration thrombectomy (Active Comparator): Aspiration thrombectomy following stent deployment and prior to removal of distal embolic protection
  Interventions: Device: Emboshield NAV6® embolic protection system (Abbott Vascular, Santa Clara, CA)

INTERVENTIONS:
Device: Emboshield NAV6® embolic protection system (Abbott Vascular, Santa Clara, CA) — Standard of care use of an embolic protection device
  Arms: Distal Embolic Protection Only
Device: Emboshield NAV6® embolic protection system (Abbott Vascular, Santa Clara, CA) — Aspiration thrombectomy following stent deployment and prior to embolic protection device removal
  Arms: Distal embolic protection and aspiration thrombectomy

SUMMARY:
The purpose of this study is to determine whether aspiration thrombectomy following carotid stent deployment will reduce the number of procedure related signals as identified by diffusion weighted MRI of the brain.

DETAILED DESCRIPTION:
Studies have demonstrated that carotid artery stenting is a safe and effective alternative to carotid endarterectomy for high or standard risk patients with symptomatic stenosis. Despite the routine use of embolic protection devices, numerous studies have shown that carotid stenting is associated with a higher degree of intracranial emboli by diffusion-weighted MRI of the brain. A potential solution to minimize this effect is the use of aspiration prior to distal embolic protection removal.

ELIGIBILITY:
Inclusion Criteria:

* ICA stenosis greater than 50 percent by carotid angiography
* Documented hemispheric ischemic stroke, TIA, amaurosis fugax, or retinal stroke in the last six months ipsilateral to the stented lesion

Exclusion Criteria:

* Subject less than 40 years of age
* Pregnant subjects
* Asymptomatic carotid stenosis
* Total occlusion of target carotid artery
* Inability to deploy distal protection device or stent in target vessel
* Allergy to both aspirin and approved thienopyridine anti-platelet drugs (clopidogrel/ticlopidine)
* Multiple carotid stenoses in same vessel that cannot be covered by single stent
* Ipsilateral intracranial stenosis requiring treatment
* Isolated common carotid stenosis
* Stenosis less than 50 percent by angiography
* Chronic or paroxysmal atrial fibrillation not treated with warfarin or dabigatran.
* Life expectancy less than 30 days
* Active bleeding diathesis
* Suspected Myocardial Infarction within 72 hours prior to carotid stenting
* Presence of intracranial tumor arteriovenous malformations or aneurysm requiring treatment
* Inability to undergo DWMRI
* Unwillingness to participate or provide consent
* Subjects using a legally authorized representative for consent for participation
* Concurrently enrolled in another study
* Stroke, TIA, amaurosis fugax ipsilateral to the treated lesion more than 6 months from randomization
* Occlusive or critical ilio-femoral disease that precludes safe femoral access to the aortic arch
* Severe atherosclerosis of the aortic arch or origin of the innominate or common carotid arteries
* Prior large stroke, multiple lacunar infarcts, or dementia
* Stenosis that contain visible thrombus

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of new, ischemic foci | 18-48 hours post procedure
  Foci of restricted diffusion will be classified by their number, location, and size

SECONDARY OUTCOMES:
Ischemic zone area | 18-48 hours post stenting
  Maximum size of new, ipsilateral,ischemic foci on post-carotid stenting diffusion-weighted MRI of the brain

CONTACTS AND LOCATIONS:
Overall Officials: James Joye, DO, Principal Investigator — Fogarty Clinical Research Inc.
Locations (2):
- United States (2):
  - El Camino Hospital, Mountain View, California
  - Northern Michigan Regional Hospital, Petoskey, Michigan